CLINICAL TRIAL: NCT01899846
Title: A Multi-Center, Non-Randomized Pharmacokinetic Study of Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL) and Its Metabolites in Blood of Women With a Singleton Pregnancy and a Previous Singleton Spontaneous Preterm Delivery
Brief Title: Pharmacokinetic Study of Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL) and Its Metabolites in Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lumara Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: HPC-PK-005
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Pregnancy
Keywords: Makena; Pharmacokinetics; Prior preterm delivery; Hydroxyprogesterone Caproate; 17P
MeSH Terms: interventions — 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Hydroxyprogesterone caproate 250 mg/ml. Detailed pharmacokinetic evaluation following first dose
  Interventions: Drug: Hydroxyprogesterone caproate 250 mg/ml
- Cohort 2 (Experimental): Hydroxyprogesterone caproate 250 mg/ml. Detailed pharmacokinetic evaluation 24 - 28 weeks gestation
  Interventions: Drug: Hydroxyprogesterone caproate 250 mg/ml
- Cohort 3 (Experimental): Hydroxyprogesterone caproate 250 mg/ml. Detailed pharmacokinetic evaluation 32 - 36 weeks gestation
  Interventions: Drug: Hydroxyprogesterone caproate 250 mg/ml

INTERVENTIONS:
Drug: Hydroxyprogesterone caproate 250 mg/ml
  Other Names: Makena; 17P

SUMMARY:
This study will evaluate the levels of hydroxyprogesterone caproate and it's metabolites in blood throughout pregnancy

There will be 3 cohorts of subjects

Cohort 1 (6 subjects) will have daily blood draws in the morning at approximately the same time each day for one week following their first dose of Makena and will have blood drawn immediately prior to 2 successive Makena doses during Epoch 1 (24 - 28 weeks) and Epoch 2 (32 - 36 weeks)

Cohort 2 (8 subjects) will have blood drawn to determine the trough concentration 7 days after their first dose of Makena. Subjects will have daily blood draws for one week following a dose of Makena given in Epoch 1 (24 - 28 weeks) and blood drawn immediately prior to 2 successive doses during Epoch 2 (32 - 36 weeks)

Cohort 3 (16 subjects) will have blood drawn to determine the trough concentration 7 days after their first dose of Makena. Subjects will have blood drawn immediately prior to 2 successive doses in Epoch 1 (24 - 28 weeks) and daily blood draws for one week following a dose of Makena given during Epoch 2 (32 - 36 weeks)

A maximum of 10 subjects will be monitored on selected days following a completed course of Makena therapy to determine the terminal elimination phase.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Singleton gestation.
* Gestational age 16 weeks 0 days to 20 weeks 6 days.
* Previous singleton spontaneous preterm delivery

Exclusion Criteria:

* Multifetal gestation.
* Known major fetal anomaly or fetal demise.
* Progestin treatment in any form in the 4 weeks prior to study entry.
* Heparin therapy during current pregnancy or history of thromboembolic disease.
* Maternal medical/obstetrical complications including hypertension requiring medication or seizure disorder.
* uterine anomaly other than fibroids
* Known hypersensitivity to hydroxyprogesterone caproate injection or its components.
* Any significant medical disorder that, in the opinion of the investigator, would be a contraindication to the use of the drug or would preclude accurate evaluation of the subject's condition or outcome or compromise the subject's safety in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of hydroxyprogesterone caproate and metabolites | First dose, 24 - 28 weeks gestation, 32 - 36 weeks gestation

SECONDARY OUTCOMES:
Plasma concentrations of hydroxyprogesterone caproate and metabolites | Up to 28 days following last dose given in week 36

CONTACTS AND LOCATIONS:
Overall Officials: Robert Birch, PhD, Study Director — Lumara Health, Inc.
Locations (6):
- United States (6):
  - Altus Research, Inc., Lake Worth, Florida
  - Rosemark WomenCare Specialists, Idaho Falls, Idaho
  - Northwestern University Department of Obstetrics and Gynecology, Chicago, Illinois
  - University of North Carolina at Chapel Hill Hospital, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - The University of Wisconsin, Madison, Wisconsin